CLINICAL TRIAL: NCT03262961
Title: Use of Sildenafil Citrate in Management of Mild Pre-eclampsia: A Randomized Controlled Trial
Brief Title: Use of Sildenafil Citrate in Management of Mild Pre-eclampsia
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Fady Nasef Tous Abdallah, Resident of Obstetrics and Gynecology Department - Assiut University, Assiut University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: assiutu252
Record Dates: First submitted 2017-08-19; First posted 2017-08-28 (Actual); Last update posted 2017-08-28 (Actual); Status verified 2017-08

CONDITIONS: Pre-Eclampsia; Mild
Keywords: Mild pre-eclampsia Sildenafil Citrate
MeSH Terms: conditions — Pre-Eclampsia; Lymphoma, Follicular | interventions — Sildenafil Citrate

STUDY DESIGN:
Intervention Model Description: - Double blinded, randomized, placebo-controlled trial.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: - It's a double blinded, randomized, placebo-controlled trial.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention Group (Active Comparator): • The intervention group will be supplied with Sildenafil Citrate (Respatio® 20mg tablets manufactured by Pharma Right Group , Egypt) according to the patient's weight by the rate of (1.5 mg/kg/day) divided into three doses per day ( every 8 hours) till termination of pregnancy.
  Interventions: Drug: Sildenafil 20 MG
- Control Group (Placebo Comparator): - The control group will be supplied with a placebo drug that has the same shape, size and color but without the active ingredient and it would also be taken in a similar way. The placebo tablet will be manufactured at the faculty of pharmacy, Assiut University.
  Interventions: Drug: Placebo Oral Tablet

INTERVENTIONS:
Drug: Sildenafil 20 MG
  Other Names: Sildenafil Citrate 20 mg ( Respatio® 20 mg)
  Arms: Intervention Group
Drug: Placebo Oral Tablet
  Other Names: Placebo drug
  Arms: Control Group

SUMMARY:
* Mild pre-eclampsia represents 75% of cases with pre-eclampsia, possible progression to severe pre-eclampsia makes mild pre-eclampsia a serious problem that requires attention.
* Previous studies have shown that expectant and conservative management of pre-eclampsia in the context of extreme prematurity may improve perinatal outcomes. Indeed, it has been estimated that for each additional day of pregnancy prolongation between 24 and 32 weeks of gestation, there is a nonlinear corresponding gain of 1% in fetal survival.
* Sildenafil citrate has been used for increasing utero-placental perfusion in cases with intrauterine growth restriction, which makes it a promising drug in management of mild pre-eclampsia.

DETAILED DESCRIPTION:
- Pre-eclampsia affects approximately 2-8% of all pregnancies worldwide. In Egypt, the prevalence of pre-eclampsia is 10.7% in a community based study. While, in hospital based studies it ranged from 9.1% to 12.5% of all deliveries. The incidence of pre-eclampsia has risen in the developing countries and even in the developed countries as the USA since the 1990s. Among the hypertensive disorders that complicate pregnancy, pre-eclampsia and eclampsia stand as major causes of maternal and perinatal morbidity and mortality worldwide. Nearly one tenth of all maternal deaths in Africa and Asia and one quarter in Latin America are associated with hypertensive diseases in pregnancy, a category that includes pre-eclampsia and the complications that are related to it.

However, the pathogenesis of pre-eclampsia is only partially understood and it is related to disturbances in placentation at the beginning of pregnancy, followed by generalized inflammation and progressive endothelial damage. There are other uncertainties too: the diagnosis, screening and management of pre-eclampsia remain controversial, as does the classification and the degree of its severity.

However, it is generally accepted as published in the different journals and in the WHO recommendations that the onset of a new episode of hypertension during pregnancy (with persistent systolic blood pressure 140 mm Hg and diastolic blood pressure 90 mm Hg or more) with the occurrence of substantial proteinuria (>0.3 g/24 h or confirmation of proteinuria by semiquantitative urine dipstick analysis with a result of at least 1+) can be used as criteria for identifying pre-eclampsia.

Although pathophysiological changes (e.g. inadequate placentation) exist from very early stages of the pregnancy, hypertension and proteinuria usually become apparent in the second half of pregnancy.

Complications of pre-eclampsia can affect both the mother and the fetus. Acutely, pre-eclampsia can be complicated by eclampsia , the development of HELLP Syndrome , hemorrhagic or ischemic stroke, liver damage and dysfunction, acute kidney injury and Acute Respiratory Distress Syndrome (ARDS).

So early detection of pre-eclampsia and prevention of the occurrence of any of its complications would save the lives of many women and prevent the possible devastating maternal and neonatal outcome of pre-eclampsia, That's why we are concerned in our study with pre-eclampsia, covering the gestational age from 28 - 36 weeks.

Mild pre-eclampsia represents 75% of cases with pre-eclampsia, possible progression to severe pre-eclampsia makes mild pre-eclampsia a serious problem that requires attention.

Previous studies have shown that expectant and conservative management of pre-eclampsia in the context of extreme prematurity may improve perinatal outcomes. Indeed, it has been estimated that for each additional day of pregnancy prolongation between 24 and 32 weeks of gestation, there is a nonlinear corresponding gain of 1% in fetal survival.

Sildenafil citrate has been used for increasing utero-placental perfusion in cases with intrauterine growth restriction, which makes it a promising drug in management of mild pre-eclampsia.

Its action is similar to the action of nitric oxide, which is a potent vasodilator, especially for the venules, besides being an inhibitor of platelet aggregation. During pregnancy, nitric oxide is synthesized in in utero-placental tissues and endothelial cells, helping to maintain low vascular resistance in the utero- and fetoplacental circulations. Phosphodiesterase metabolizes cyclic guanosine monophosphate; therefore, phosphodiesterase type 5 inhibition leads to cyclic guanosine monophosphate increase with associated vasodilation, independently of nitric oxide. Therefore, phosphodiesterase type 5 inhibitors have the potential to achieve similar therapeutic goals when compared with nitric oxide.

A potential advantage of phosphodiesterase type 5 inhibitors is that they may overcome the main limitation to nitric oxide use in pregnancy, which is tolerance and headaches. The most studied phosphodiesterase type 5 inhibitor is sildenafil citrate, which has previously shown promising outcomes both in vitro and in animal studies.

That is why we decided to study the role of Sildenafil Citrate in expectant and conservative management of mild pre-eclampsia, as it has shown its ability to be beneficial to both the mother and the fetus through increasing the maternofetal circulation perfusion and achieving a maternal hemodynamic stability and compare it to the current NICE (National Institute for Health and Care Excellence) guidelines that are currently used, that recommends conservative management of mild pre-eclampsia through control of maternal blood pressure and frequent screening of maternal laboratory investigations' abnormalities to detect possible progression to severe pre-eclamptic toxemia.

ELIGIBILITY:
Inclusion Criteria:

1. Uncomplicated mild pre-eclampsia; No clinical or investigatory findings suggestive severe pre-eclamptic toxemia.
2. Gestational age of 28 - 36 weeks by good dates according to ACOG's - committee on obstetric practice - Method for Estimating Due Date (2014) who will receive the study's drug for at least one week before termination.
3. Singleton viable pregnancy.
4. Age: 18-35 years.

Exclusion Criteria:

1. Severe pre-eclamptic toxemia (according to the NICE guidelines (2010): Hypertension in pregnancy: diagnosis and management)
2. Intrauterine growth retardation.
3. Use of medication that could interact with sildenafil citrate such as nitrates erythromycin, ketoconazole, itraconazole, antiretroviral agents and others.
4. Presence of maternal co-morbidity disease as: DM, chronic hypertension, congestive heart failure, chronic kidney disease and SLE.
5. Placenta previa.
6. The patient is using aspirin.
7. The presence of a contraindication to the use of sildenafil citrate:

   * Hypersensitivity to sildenafil citrate or any of the tablet ingredients.
   * Patients with severe cardiovascular disease such as established cardiac failure and unstable angina pectoris.
   * Previous episode of non-arteritic anterior ischaemic optic neuropathy.
   * Severe hepatic impairment.
   * Hypotension (blood pressure <90/50 mmHg).
   * Hypertension (blood pressure >170/110 mmHg).
   * Recent history of stroke or myocardial infarction.
   * Known hereditary degenerative retinal disorders such as retinitis pigmentosa.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Pregnant females
Enrollment: 80 (Estimated)
Dates: Start 2016-09-15 (Actual); Primary Completion 2017-12-15 (Estimated); Study Completion 2018-01-15 (Estimated)

PRIMARY OUTCOMES:
Gestational age at time of termination and maternal outcome. | up to 37 weeks of gestation
  Gestational age at time of termination and maternal outcome in terms of whether the disease would progress to severe pre-eclampsia or not.

SECONDARY OUTCOMES:
Neonatal outcome. | up to 37 weeks of gestation
  Neonatal outcome in terms of survival and neonatal well-being ( by obtaining the birth weight and the apgar score at 1 and 5 minutes and direct postnatal need to NICU).
Control of maternal blood pressure. | up to 37 weeks of gestation
  Control of maternal blood pressure.
Method of termination of pregnancy. | up to 37 weeks of gestation
  Method of termination of pregnancy.
Identification of the side effects from the use of sildenafil citrate. | up to 37 weeks of gestation
  Identification of possible maternal side effects from the use of sildenafil citrate i.e.; headache, flushing and dyspepsia.
Evaluation of the effect of sildenafil citrate on the feto-maternal circulation through the Doppler ultrasound. | up to 37 weeks of gestation
  Evaluation of the effect of sildenafil citrate on the feto-maternal circulation through the Doppler ultrasound.

CONTACTS AND LOCATIONS:
Overall Officials: Fady Abdallah, Principal Investigator — Assiut University; Hasan Kamel, Study Director — Assiut University; Hisham Abou-Taleb, Study Director — Assiut University
Locations (1):
- Assiut Univeristy Hospitals, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Eiland E, Nzerue C, Faulkner M. Preeclampsia 2012. J Pregnancy. 2012;2012:586578. doi: 10.1155/2012/586578. Epub 2012 Jul 11. PMID 22848831
- [Background] El-Moselhy, E; Khalifa, H; Amer, S (2011). "Risk Factors and Impacts of Pre-Eclampsia: An Epidemiological Study among Pregnant Mothers in Cairo, Egypt" J Am Sci 7(5): 311-323.
- [Background] Steegers EA, von Dadelszen P, Duvekot JJ, Pijnenborg R. Pre-eclampsia. Lancet. 2010 Aug 21;376(9741):631-44. doi: 10.1016/S0140-6736(10)60279-6. Epub 2010 Jul 2. PMID 20598363
- [Background] Khan KS, Wojdyla D, Say L, Gulmezoglu AM, Van Look PF. WHO analysis of causes of maternal death: a systematic review. Lancet. 2006 Apr 1;367(9516):1066-1074. doi: 10.1016/S0140-6736(06)68397-9. PMID 16581405
- [Background] Campbell OM, Graham WJ; Lancet Maternal Survival Series steering group. Strategies for reducing maternal mortality: getting on with what works. Lancet. 2006 Oct 7;368(9543):1284-99. doi: 10.1016/S0140-6736(06)69381-1. PMID 17027735
- [Background] Roberts JM, Cooper DW. Pathogenesis and genetics of pre-eclampsia. Lancet. 2001 Jan 6;357(9249):53-6. doi: 10.1016/s0140-6736(00)03577-7. PMID 11197372
- [Background] Arulkumaran N, Lightstone L. Severe pre-eclampsia and hypertensive crises. Best Pract Res Clin Obstet Gynaecol. 2013 Dec;27(6):877-84. doi: 10.1016/j.bpobgyn.2013.07.003. Epub 2013 Aug 17. PMID 23962474
- [Background] Mustafa R, Ahmed S, Gupta A, Venuto RC. A comprehensive review of hypertension in pregnancy. J Pregnancy. 2012;2012:105918. doi: 10.1155/2012/105918. Epub 2012 May 23. PMID 22685661
- [Background] Report of the National High Blood Pressure Education Program Working Group on High Blood Pressure in Pregnancy. Am J Obstet Gynecol. 2000 Jul;183(1):S1-S22. PMID 10920346
- [Background] Sibai BM. Magnesium sulfate prophylaxis in preeclampsia: Lessons learned from recent trials. Am J Obstet Gynecol. 2004 Jun;190(6):1520-6. doi: 10.1016/j.ajog.2003.12.057. PMID 15284724
- [Background] Hypertension in pregnancy. Report of the American College of Obstetricians and Gynecologists' Task Force on Hypertension in Pregnancy. Obstet Gynecol. 2013 Nov;122(5):1122-1131. doi: 10.1097/01.AOG.0000437382.03963.88. No abstract available. PMID 24150027
- [Background] Sibai BM, Mercer BM, Schiff E, Friedman SA. Aggressive versus expectant management of severe preeclampsia at 28 to 32 weeks' gestation: a randomized controlled trial. Am J Obstet Gynecol. 1994 Sep;171(3):818-22. doi: 10.1016/0002-9378(94)90104-x. PMID 8092235
- [Background] Haddad B, Deis S, Goffinet F, Paniel BJ, Cabrol D, Siba BM. Maternal and perinatal outcomes during expectant management of 239 severe preeclamptic women between 24 and 33 weeks' gestation. Am J Obstet Gynecol. 2004 Jun;190(6):1590-5; discussion 1595-7. doi: 10.1016/j.ajog.2004.03.050. PMID 15284743
- [Background] Manktelow BN, Seaton SE, Field DJ, Draper ES. Population-based estimates of in-unit survival for very preterm infants. Pediatrics. 2013 Feb;131(2):e425-32. doi: 10.1542/peds.2012-2189. Epub 2013 Jan 14. PMID 23319523
- [Background] Cauli O, Herraiz S, Pellicer B, Pellicer A, Felipo V. Treatment with sildenafil prevents impairment of learning in rats born to pre-eclamptic mothers. Neuroscience. 2010 Dec 1;171(2):506-12. doi: 10.1016/j.neuroscience.2010.08.065. Epub 2010 Sep 9. PMID 20832451
- [Background] Coppage KH, Sun X, Baker RS, Clark KE. Expression of phosphodiesterase 5 in maternal and fetal sheep. Am J Obstet Gynecol. 2005 Sep;193(3 Pt 2):1005-10. doi: 10.1016/j.ajog.2005.05.054. PMID 16157102
- [Background] Samangaya RA, Mires G, Shennan A, Skillern L, Howe D, McLeod A, Baker PN. A randomised, double-blinded, placebo-controlled study of the phosphodiesterase type 5 inhibitor sildenafil for the treatment of preeclampsia. Hypertens Pregnancy. 2009 Aug;28(4):369-82. doi: 10.3109/10641950802601278. PMID 19843000
- [Background] Trapani A Jr, Goncalves LF, Trapani TF, Franco MJ, Galluzzo RN, Pires MM. Comparison between transdermal nitroglycerin and sildenafil citrate in intrauterine growth restriction: effects on uterine, umbilical and fetal middle cerebral artery pulsatility indices. Ultrasound Obstet Gynecol. 2016 Jul;48(1):61-5. doi: 10.1002/uog.15673. PMID 26279411
- [Background] Galie N, Ghofrani HA, Torbicki A, Barst RJ, Rubin LJ, Badesch D, Fleming T, Parpia T, Burgess G, Branzi A, Grimminger F, Kurzyna M, Simonneau G; Sildenafil Use in Pulmonary Arterial Hypertension (SUPER) Study Group. Sildenafil citrate therapy for pulmonary arterial hypertension. N Engl J Med. 2005 Nov 17;353(20):2148-57. doi: 10.1056/NEJMoa050010. PMID 16291984
- [Background] ACOG Practice bulletin no. 134: fetal growth restriction. Obstet Gynecol. 2013 May;121(5):1122-1133. doi: 10.1097/01.AOG.0000429658.85846.f9. PMID 23635765
- [Background] Matt H, Nigel J. (2016) "Renal disease in pregnancy" ;Obstet Gynaecol Reprod Med; 26:46-52
- [Result] Dastjerdi MV, Hosseini S, Bayani L. Sildenafil citrate and uteroplacental perfusion in fetal growth restriction. J Res Med Sci. 2012 Jul;17(7):632-6. PMID 23798922
- [Result] McKeeman GC, Ardill JE, Caldwell CM, Hunter AJ, McClure N. Soluble vascular endothelial growth factor receptor-1 (sFlt-1) is increased throughout gestation in patients who have preeclampsia develop. Am J Obstet Gynecol. 2004 Oct;191(4):1240-6. doi: 10.1016/j.ajog.2004.03.004. PMID 15507947
- [Result] Moncada S, Higgs A. The L-arginine-nitric oxide pathway. N Engl J Med. 1993 Dec 30;329(27):2002-12. doi: 10.1056/NEJM199312303292706. No abstract available. PMID 7504210
- [Result] Learmont JG, Poston L. Nitric oxide is involved in flow-induced dilation of isolated human small fetoplacental arteries. Am J Obstet Gynecol. 1996 Feb;174(2):583-8. doi: 10.1016/s0002-9378(96)70432-5. PMID 8623789
- [Result] Lees C, Valensise H, Black R, Harrington K, Byiers S, Romanini C, Campbell S. The efficacy and fetal-maternal cardiovascular effects of transdermal glyceryl trinitrate in the prophylaxis of pre-eclampsia and its complications: a randomized double-blind placebo-controlled trial. Ultrasound Obstet Gynecol. 1998 Nov;12(5):334-8. doi: 10.1046/j.1469-0705.1998.12050334.x. PMID 9819872
- [Result] Trapani A Jr, Goncalves LF, Pires MM. Transdermal nitroglycerin in patients with severe pre-eclampsia with placental insufficiency: effect on uterine, umbilical and fetal middle cerebral artery resistance indices. Ultrasound Obstet Gynecol. 2011 Oct;38(4):389-94. doi: 10.1002/uog.8983. PMID 21374750
- [Result] Wareing M, Myers JE, O'Hara M, Baker PN. Sildenafil citrate (Viagra) enhances vasodilatation in fetal growth restriction. J Clin Endocrinol Metab. 2005 May;90(5):2550-5. doi: 10.1210/jc.2004-1831. Epub 2005 Feb 15. PMID 15713717
- [Result] Trapani A Jr, Goncalves LF, Trapani TF, Vieira S, Pires M, Pires MMS. Perinatal and Hemodynamic Evaluation of Sildenafil Citrate for Preeclampsia Treatment: A Randomized Controlled Trial. Obstet Gynecol. 2016 Aug;128(2):253-259. doi: 10.1097/AOG.0000000000001518. PMID 27400005

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-09-01): https://cdn.clinicaltrials.gov/large-docs/61/NCT03262961/Prot_SAP_000.pdf